CLINICAL TRIAL: NCT06555627
Title: Project EMBRACE: Embracing Morning BReakfast and Activity for Classroom Engagement
Brief Title: Embracing Morning BReakfast and Activity for Classroom Engagement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: 2024-0746
Record Dates: First submitted 2024-07-29; First posted 2024-08-15 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Child Development

STUDY DESIGN:
Intervention Model Description: 2x2 factorial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise and High Protein Breakfast (Experimental): Children in this group will be given given breakfast each morning at 7:30 am and participate in a 30-minute bout of physically active games of moderate to vigorous intensity at 8 am.
  Nutrition Intervention. For 5 days children will receive a high protein breakfast comprised of baked items (i.e. waffles with syrup) and Greek yogurt. The high protein meal will aim for 40% protein, 40% carbohydrates, and 20% fat. Meals will be served with a cup of water.
  Exercise Intervention. For 5 days, a 30-min physical activity bout including a 5-minute warm up and cool down will be provided to participants in this group. The aim is for students to achieve an average heart rate above 150 for the session, not including warm up or cool down. To monitor intensity, the participant will wear heart rate monitors around their chest and waist-worn accelerometers
  Interventions: Behavioral: High Protein Breakfast; Behavioral: Morning Exercise
- High Protein Breakfast Only (Active Comparator): Nutrition Intervention. For 5 days children will receive a high protein breakfast comprised of baked items (i.e. waffles with syrup) and Greek yogurt. The high protein meal will aim for 40% protein, 40% carbohydrates, and 20% fat. Meals will be served with a cup of water.
  Interventions: Behavioral: High Protein Breakfast
- Exercise and High Carb Breakfast (Active Comparator): Exercise Intervention. For 5 days, a 30-min physical activity bout including a 5-minute warm up and cool down will be provided to participants in this group. The aim is for students to achieve an average heart rate above 150 for the session, not including warm up or cool down. To monitor intensity, the participant will wear heart rate monitors around their chest and waist-worn accelerometers.
  For 5 days children will receive a high carb breakfast that will be comprised of 15% protein, 65% carbohydrates and 20% fat. Total energy content, fat, sugar, fiber, energy density, are similar between the breakfast meals.
  Interventions: Behavioral: Morning Exercise; Behavioral: High Carb Breakfast
- High Carb Breakfast Only (Placebo Comparator): For 5 days children will receive a high carb breakfast that will be comprised of 15% protein, 65% carbohydrates and 20% fat. Total energy content, fat, sugar, fiber, energy density, are similar between the breakfast meals.
  Interventions: Behavioral: High Carb Breakfast

INTERVENTIONS:
Behavioral: High Protein Breakfast — For 5 days children will receive a high protein breakfast comprised of baked items (i.e. waffles with syrup) and Greek yogurt. The high protein meal will aim for 40% protein, 40% carbohydrates, and 20% fat. Meals will be served with a cup of water.
  Arms: Exercise and High Protein Breakfast; High Protein Breakfast Only
Behavioral: Morning Exercise — Exercise Intervention. For 5 days, a 30-min physical activity bout including a 5-minute warm up and cool down will be provided to participants in this group. The aim is for students to achieve an average heart rate above 150 for the session, not including warm up or cool down. To monitor intensity, the participant will wear heart rate monitors around their chest and waist-worn accelerometers.
  Arms: Exercise and High Carb Breakfast; Exercise and High Protein Breakfast
Behavioral: High Carb Breakfast — For 5 days children will receive a high carb breakfast that will be comprised of 15% protein, 65% carbohydrates and 20% fat. Total energy content, fat, sugar, fiber, energy density, are similar between the breakfast meals.
  Arms: Exercise and High Carb Breakfast; High Carb Breakfast Only

SUMMARY:
This experiment will test the effects of healthy breakfast and morning exercise on children's focus and classroom behavior. Food and exercise each influence child focus, but little is known about their effects on classroom behavior and less about their combined effects. For one week (Monday-Friday), 10 children will be randomly assigned to receive healthy breakfast and morning exercise, 10 assigned to only healthy breakfast, 10 to only exercise, and 10 to neither. After exercise and breakfast, study staff will assess how focused children are during class-time, ask them to complete puzzle-like tasks, and wear a helmet that measures brain blood flow

DETAILED DESCRIPTION:
Specific Aims:

Specific Aim 1: Determine the independent and convergent effects of breakfast and exercise on child classroom behavior using systematic classroom observations.

Hypothesis 1: Groups assigned to receive protein-rich breakfast (1 & 3) will demonstrate greater engagement and reduced off-task behavior compared with those receiving high carb breakfast (groups 2 & 4) (the main effect of high-protein breakfast). Groups receiving morning exercise (2 & 3) will demonstrate great engagement and reduced off-task behavior compared with groups not receiving exercise (1 & 4) (main effect of exercise). Children receiving both exercise and breakfast (group 3), will demonstrate greater improvements than those receiving just one (1 vs. 3 & 2 vs. 3), the interaction effect.

Specific Aim 2: Determine the independent and convergent effects of breakfast and physical activity on inhibitory control and attention using computerized executive function tasks.

Hypothesis 2: It is hypothesized that our data will show a main effect of protein rich breakfast on neuropsychological task performance (groups 1 & 3 vs. groups 2 & 4), a main effect of morning exercise (2 & 3 vs. 1 & 4), and an interaction effect favoring the combination of breakfast and exercise beyond either in isolation (3 vs. 1, 3 vs. 2).

Specific Aim 3: Explore potential changes in brain activity by assessing blood flow via functional near-infrared spectroscopy (fNIRS) in the prefrontal cortex, while completing the computerized cognitive tasks.

Hypothesis 3: Results are expected to evidence similar patterns as aims 1 and 2, such that blood flow in the prefrontal cortex, will increase more in groups receiving both, relative to those receiving just one, and those receiving neither. Relationships between cerebral blood flow, task performance, and classroom behavior will be assessed.

Background:

Strong experimental and observational evidence supports connections between nutrition, physical activity, and neurocognitive development. In fact, one of the first interventions to show that exercise improves cognitive abilities in elementary-aged children was conducted at the University of Illinois Urbana Champaign, and several subsequent studies have replicated these results. Many studies assessing diet quality indicate a clear link between diet quality and cognition in children. While these outcomes are important for researchers, their perceived importance to parents and teachers lies in their promise to influence academic outcomes. For example, exercise improves cognitive inhibition on lab-based tasks, but teachers want to see that the benefit generalizes to raising their hands before speaking. Here, there is surprisingly little data, limiting adoption of interventions.

Another consideration regarding health behaviors is socioeconomic status, as individuals from low income neighborhoods as well as racial/ethnic minorities have shown to have poorer dietary patterns, lower rates of physical activity, and higher rates of obesity, making children in these groups particularly vulnerable to falling behind in academic achievement and cognitive development. Thus, interventions to improve such health behaviors ought to target children representing these populations as they likely have the most gain from healthy lifestyle changes.

Finally, interventions conducted in schools are particularly advantageous as children spend most of their day in schools not only during instruction but also before and after school as childcare while parents are working. Lastly, while many observational and experimental studies show clear diet-cognition and exercise-cognition interactions, these are almost always studied in isolation without examining combined effects. Which is most important? How much benefit does the combination of diet and exercise provide above and beyond either in isolation?

The outcomes of interest include children's classroom behavior, specifically time spent on and off task, behavioral cognitive skills such as accuracy and reaction time on computerized tasks assessing attention and inhibitory control, and blood flow to specific areas of the brain associated with attention and classroom behavior. This pilot study will implement a 1-week (Monday-Friday) school-based intervention using a 2 x 2 factorial design with 2 factors, morning exercise (yes/no) and breakfast (protein rich/carb rich) and 2 levels of each factor (yes or no). Children will be randomized into one of four intervention groups, 1) protein rich breakfast only, 2) exercise and carb rich breakfast, 3) both protein rich breakfast and exercise, and 4) carb rich breakfast only. Monday, Wednesday, and Friday of that week, children's classroom behavior will be monitored via a recording on a camera placed in their classroom. Friday afternoon children's cognitive function and brain blood flow will be assessed. Randomization will be conducted post baseline by a study co-investigator, Dr. Naiman Kahn using a block randomization scheme which will be applied during each wave. Waves will be in sizes that are divisible by four. Data collectors will be blind to condition. Interventions will not collect data.

The current study is a school based intervention. Children will be monitored for one week prior to intervention implementation in order to provide baseline assessments of classroom behavior, cognition, and brain blood flow. The intervention will be implemented the following week and post testing will occur during the same week on Monday, Wednesday, and Friday. Following completion of the study, all participants will be offered five days of breakfast and five days of morning exercise regardless of group assignment.

The following procedure will be followed:

Parent's will complete a demographics survey after consent to confirm the participants, age, biological sex, date of birth, race/ethnicity, household income/educational status, and any diagnosis of neuropsychological disorders such as autism spectrum disorder or Attention-Deficit Hyperactivity/Impulsivity Disorder (ADHD).

Baseline Testing: For one week prior to the intervention, children's classroom behavior will be observed three times during the week (Monday-Friday) using the Behavioral Observation of Students in Schools (BOSS) systematic observation tool. Further, baseline brain function via Functional Near Infrared Spectroscopy (fNIRS) and cognitive testing via performance on computerized tasks will be assessed at the end of the week on Friday along with height and weight.

Aerobic fitness will be assessed via a shuttle run. This test allows for a group assessment of aerobic fitness by instructing children to run in sync with a series of beeps for 20 meters. The frequency of the beeps gradually increases, requiring participants to run faster each round. Once a child cannot keep up with the pace, the test is completed. This assessment will only be completed once at baseline.

During morning physical activity sessions hart rate will be recorded using the first beat heart rate system, which includes chest straps. For the entire baseline week, children will be asked to wear an accelerometer on their hip to assess their physical activity level throughout the day. Children's height and weight will be assessed once at baseline using a scale and stadiometer.

ELIGIBILITY:
Inclusion Criteria:

* 6-11 years old
* Enrolled at the participating school

Exclusion Criteria:

* Younger than 5 years old
* Older than 12 years old
* Not enrolled in a participating school
* Allergic to dairy or gluten

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Behavioral Observation of Students in Schools (BOSS) - Classroom Engagement (Shapiro et al., 2003) | Classroom observations will occur between 9:00am and 11:30am on 3 days during the baseline week and on 3 days during the intervention week.
  The Behavioral Observation of Students in Schools (BOSS) (Shapiro et al., 2003) is a systematic observation tool that assesses children's classroom behavior, including active and passive engagement, and the frequency of three kinds of off-task behavior: motor, verbal, and passive. The primary outcome in this study will be engaged time during instruction this will add up actively and passively engaged time and be represented by the percentage of time during instruction that students are engaged in instruction. The BOSS provides the percentage of observation intervals during which children are engaged in instruction (0%-100%) and a higher percentage is better.

SECONDARY OUTCOMES:
Behavioral Observation of Students in Schools (BOSS) - Off-Task Motor (Shapiro et al., 2003) | Classroom observations will occur between 9:00am and 11:30am on 3 days during the baseline week and on 3 days during the intervention week.
  The Behavioral Observation of Students in Schools (BOSS) (Shapiro et al., 2003) is a systematic observation tool that assesses children's classroom behavior, including active and passive engagement, and the frequency of three kinds of off-task behavior: motor, verbal, and passive. The primary outcome in this study will be engaged time during instruction this will add up actively and passively engaged time and be represented by the percentage of time during instruction that students are engaged in instruction. The BOSS provides the percentage of observed intervals during which children are off-task motor during instruction (0%-100%) and a lower percentage is better.
Behavioral Observation of Students in Schools (BOSS) - Off-Task Verbal (Shapiro et al., 2003) | Classroom observations will occur between 9:00am and 11:30am on 3 days during the baseline week and on 3 days during the intervention week.
  The Behavioral Observation of Students in Schools (BOSS) (Shapiro et al., 2003) is a systematic observation tool that assesses children's classroom behavior, including active and passive engagement, and the frequency of three kinds of off-task behavior: motor, verbal, and passive. The primary outcome in this study will be engaged time during instruction this will add up actively and passively engaged time and be represented by the percentage of time during instruction that students are engaged in instruction. The BOSS provides the percentage of observed intervals during which children are off-task verbal during instruction (0%-100%) and a lower percentage is better.
Behavioral Observation of Students in Schools (BOSS) - Off-Task Passive (Shapiro et al., 2003) | Classroom observations will occur between 9:00am and 11:30am on 3 days during the baseline week and on 3 days during the intervention week.
  The Behavioral Observation of Students in Schools (BOSS) (Shapiro et al., 2003) is a systematic observation tool that assesses children's classroom behavior, including active and passive engagement, and the frequency of three kinds of off-task behavior: motor, verbal, and passive. The primary outcome in this study will be engaged time during instruction this will add up actively and passively engaged time and be represented by the percentage of time during instruction that students are engaged in instruction. The BOSS provides the percentage of observed intervals during which children are off-task passive during instruction (0%-100%) and a lower percentage is better.
Neurocognitive inhibition test - Fishy Flanker Test | Neurocognitive testing will occur on Friday morning between 9am and 11:30am during the baseline testing week and then again the following Friday at the same time during the intervention week
  The Fishy Flanker test requires the participant to focus on a given stimulus while inhibiting attention to stimuli flanking it. In this version of the task, younger participants see a picture of a fish flanked by two other fish on either side. On congruent trials, all the fish are pointing in the same direction. The flanker provides both an accuracy score (0%-100%) and a reaction time score in milliseconds. Higher accuracy and lower time in ms are considered better.
Neurocognitive inhibition test - Go/No-go | Neurocognitive testing will occur on Friday morning between 9am and 11:30am during the baseline testing week and then again the following Friday at the same time during the intervention week
  The Go/No-go task is a simple experimental paradigm that requires participants to respond by pressing a button when they see a "go" signal, and not respond when they see the "no-go" signal. The key behavior measured with this experiment is the participants' ability to withhold a response on No-go trials. The Go/No-Go provides both an accuracy score (0%-100%) and a reaction time score in milliseconds. Higher accuracy and lower time in ms are considered better.
Brain blood flow as assessed by functional near infrared spectroscopy (fNIRS) | Neurocognitive testing, including fNIRS will occur on Friday morning between 9am and 11:30am during the baseline testing week and then again the following Friday at the same time during the intervention week
  Functional near-infrared spectroscopy (fNIRS) is an emerging hemodynamic neuroimaging brain-computer interface (BCI) technology that indirectly measures neuronal activity in the brain's cortex via neuro-vascular coupling. The fNIRS outcomes include levels of oxyhemoglobin and deoxyhemoglobin. These measurements approximately equate to the blood-oxygen-level dependent (BOLD) signal measured in functional magnetic resonance imaging (fMRI). The results are interpreted together with the cognitive performance on task.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bustamante, Principal Investigator — University of Illinois Chicago
Locations (1):
- Altus Academy, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No